CLINICAL TRIAL: NCT04254133
Title: Genetic Information to Inform Treatment and Screening (GIFTS) Study for Prostate Cancer
Brief Title: Genetic Information to Inform Treatment and Screening for Prostate Cancer, GIFTS Study
Acronym: GIFTS
Status: Enrolling by invitation | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: RG1004177; P50CA097186 (NIH); NCI-2020-00933 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 8754 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires; Specimen Handling; Genetic Testing; Genetic Counseling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Ascertainment: Men with prostate cancer
  Interventions: Behavioral: Questionnaire; Procedure: Biospecimen Collection; Diagnostic Test: Genetic Testing; Other: Genetic Counseling; Other: Laboratory Biomarker Analysis
- Family Recruitment: Male relatives of men with prostate cancer
  Interventions: Behavioral: Questionnaire; Procedure: Biospecimen Collection; Diagnostic Test: Genetic Testing; Other: Genetic Counseling; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Behavioral: Questionnaire — Complete questionnaire
  Other Names: Questionnaires
Procedure: Biospecimen Collection — Provide saliva samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Diagnostic Test: Genetic Testing — Undergo genetic testing
  Other Names: Genetic Analysis; Genetic Examination; Genetic Test
Other: Genetic Counseling — Undergo counseling
Other: Laboratory Biomarker Analysis — Correlative Studies

SUMMARY:
This trial studies the role of inherited (present at birth) mutations in cancer risk genes such as BRCA2, BRCA1, ATM, CHEK2, and others in relation to prostate cancer. This study may help researchers understand the frequency and importance of inherited mutations in cancer risk genes in patients with prostate cancer and potentially help identify better ways to treat cancer in patients who have a mutation in one of these genes.

DETAILED DESCRIPTION:
OUTLINE:

Participants complete questionnaire over 20 minutes at baseline, then undergo collection of saliva sample for genetic testing. Participants identified to have an inherited mutation in a deoxyribonucleic acid (DNA) repair gene undergo genetic counseling. Participants whose genetic testing does not indicate an inherited mutation in a DNA repair gene receive a letter thanking them for their participation and emphasizing the importance of ongoing communication with their physician and family members about cancer risk. Participants may also receive an educational flyer with or without a educational video regarding prostate cancer and genetic testing.

Participants will be sent newsletters every year to encourage study engagement and update health questionnaires every two years.

ELIGIBILITY:
Inclusion Criteria: Case Ascertainment [Cancer Surveillance System (CSS)/Washington State Cancer Registry (WSCR)]:

* Signed informed consent form providing agreement for germline genetic and molecular testing, use release of health and research information; and
* Male aged 35 to 89 years; and
* Diagnosis of prostate cancer; and
* Resident of Washington state at diagnosis; and
* Willing to complete a questionnaire (online or on paper) to provide basic demographic information, family cancer history, and health history; and
* Willing and able to provide a saliva sample; and
* United States (U.S.) mailing address.

Inclusion Criteria: Case Ascertainment [UW Medical Center (UWMC)/UW Harborview Medical Center (UWHMC)]:

* Signed informed consent form providing agreement for germline genetic and molecular testing, use release of health and research information; and
* Male aged 35 to 89 years; and
* Diagnosis of prostate cancer; and
* Self-identifies as Black, African American, or African; and
* Receiving care at UWMC or UWHMC; and
* Willing and able to provide a saliva sample; and
* Able to provide either a U.S. mailing address or Email address or Phone number.

Inclusion Criteria: Family Recruitment

* Signed informed consent form providing agreement for germline genetic and molecular testing, use and release of health and research information; and
* Males aged 35 to 89 years; and
* Willingness to complete a questionnaire (online or on paper) to provide basic demographic information, family cancer history, and health history; and
* Willing and able to provide a saliva sample; and
* U.S. mailing address

Exclusion Criteria: Case Ascertainment

* Unable to provide informed consent, e.g., decisional impairment
* Prior bone marrow transplant
* Currently under treatment for a hematologic malignancy
* Study team members

Exclusion Criteria: Family Recruitment

* Unable to provide informed consent, e.g., decisional impairment
* Prior bone marrow transplant
* Currently under treatment for a hematologic malignancy
* Study team members

Ages: 35 Years to 89 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients living in Washington State with a new diagnosis of prostate cancer and first degree relatives of patients with prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 1360 (Estimated)
Dates: Start 2018-11-30 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Identification of a population-based cohort of men with prostate cancer (PC) and germline deoxyribonucleic acid (DNA) repair gene (gDRG) mutations | From the start of study through death (up to 20 years)
  Identification to be determined through the Washington State Cancer Registry and by genetic testing on saliva samples for inherited mutations in cancer risk genes such as BRCA2, BRCA1, ATM, and others in prostate cancer.
Clinical, pathologic, and molecular predictors of gDRG mutation carriers for men with PC | From the start of study through death (up to 20 years)
  Predictors to be identified by analyzing information provided by participants on their health history and potentially further testing or chart review on participants who consent to future contact.
Utility and feasibility of cascade genetic testing through use of family history of men with PC identified to have gDRG mutations | From the start of study through death (up to 20 years)
  To be determined by collection of information about participants' family history and subsequent analysis of cascade genetic testing outcomes.
Identification of a cohort of men with gDRG mutations without PC | From the start of study through death (up to 20 years)
  Identification to be determined through family history of men with PC identified through the Washington State Cancer Registry and by genetic testing on saliva samples for inherited mutations in cancer risk genes such as BRCA2, BRCA1, ATM, and others in prostate cancer.
Effectiveness of a germline genetic testing education video: Number of participants who participate in genetic testing after watching germline genetic testing video | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Darst, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium; Heather H Cheng, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium; Daniel W Lin, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium; Colin C Pritchard, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No